CLINICAL TRIAL: NCT01807702
Title: 13C-Pyruvate Breath Test Pilot Study
Brief Title: 13C-Pyruvate Breath Test
Acronym: PBT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB# 654-10
Record Dates: First submitted 2013-02-22; First posted 2013-03-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: dichloroacetate; pyruvate; lactate; pyruvate dehydrogenase
MeSH Terms: interventions — Dichloroacetic Acid; Pyruvic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13C-pyruvate,13C-Lactate and dichloroacetate (Experimental): During the first day of the subjects participation pyruvate will be given and blood, breath and buccal cell samples will be collected over a two hour period. On the last day DCA will be given.
  Interventions: Drug: 13C-Pyruvate 13C-lactate and dichloroacetate

INTERVENTIONS:
Drug: 13C-Pyruvate 13C-lactate and dichloroacetate — Subjects will receive pyruvate and have blood,CO2, and buccal cell samples collected. The second visit the subjects will receive a dose of dichloroacetate before the pyruvate is given
  Other Names: dichloroacetate; pyruvate; CO2 collection

SUMMARY:
The purpose of the test is to measure an enzyme called pyruvate. Subjects will fast for 12 hours and then undergo a breath test, have blood drawn, and cells from the inside of the mouth collected over a 12 hour period. The tests will be repeated at least a week later and subjects receive a dose of dichloroacetate (DCA)

DETAILED DESCRIPTION:
Subjects will be screened with a history and physical and have baseline laboratory values drawn to assure that the subject is healthy.Subjects will fast for 12 hours before the test. The next day they will receive a dose of 25mg of pyruvate dissolved in 80ml of Crystal Light. The pyruvate used in this study will be prepared with a nonradioactive form of carbon, called a stable isotope. It poses no hazard to the subject's health. About 50 mls of blood will be drawn over a 120 minute time period from an IV catheter placed in the arm. Subjects will also be asked to exhale into a plastic tube about 12 times in 120 minutes to collect 13C carbon dioxide (13CO2). Cells from inside of the mouth will be collected by subjects swishing a tablespoon of mouth wash for one minute and then spitting it into a sterile plastic tube. At least one week following the first admission subjects will return to repeat the above procedure and receive 25mg of dichloroacetate (DCA) one hour before receiving the pyruvate. Then the same samples will be collected. Subjects have the option of doing the tests 4 times receiving the DCA on the last visit.

ELIGIBILITY:
Inclusion Criteria:- healthy volunteers

* normal history,
* normal physical
* normal baseline laboratory data.

Exclusion Criteria:

* Any illness
* Chronic health condition
* Use of street drugs
* Taking medication
* Abnormal labs Abnormal physical exam -

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Effect of dichloroacetate on pyruvate dehydrogenase and 13C02 production. | Baseline to one year
  Dichloroacetate is an activator of pyruvate dehydrogenase (PDH). It will be administered to the patient who will then undergo the pyruvate breath test to measure the amount of 13CO2 expressed. The activity of 13CO2 as measured by a concentration curve will reflect PDH activity.

SECONDARY OUTCOMES:
Blood Lactate levels and 13CO2 Response to DCA | Baseline to one year
  There will be a correlation between blood lactate levels and 13CO2 in response to DCA administration by comparing CO2 breath peaks in the concentration curve compared to serum lactate levels for same time period.
Conversion of 13C pyruvate to 13C pyruvate | Baseline to One Year
  There will be no reduction in the conversion of 13C-pyruvate to 13C-lactate in blood in response to DCA administration.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States